CLINICAL TRIAL: NCT05279274
Title: ShorT Stay Aneurysm Repair (STAR): A 23-hour Endovascular Abdominal Aortic Aneurysm Repair Pathway With Evaluation of Eligibility, Uptake, Viability, Acceptability, Safety and Cost
Brief Title: ShorT Stay Aneurysm Repair Study
Acronym: STAR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Collaborators: W.L.Gore & Associates (Industry); Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 21SM7261; IRAS 302827 (Other: The Health Research Authority (HRA))
Record Dates: First submitted 2022-03-03; First posted 2022-03-15 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Abdominal Aortic Aneurysm Without Rupture
Keywords: Abdominal aortic aneurysm; Day case; Endovascular aneurysm repair; Short stay
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective observational cohort study to assess the eligibility, uptake, viability, acceptability, safety, and cost of a ShorT stay (23-hour) Aneurysm Repair (STAR) pathway. Outcomes will be collected for up to 1 year.

DETAILED DESCRIPTION:
The STAR study is a prospective multicentre observational cohort study to assess the eligibility, uptake, viability, acceptability, safety, and cost of a short stay (23-hour) aneurysm pathway for infrarenal AAA patients.

The study will take place at least at five sites in the United Kingdom. Over a 12-month recruitment period, all patients with AAA referred to or diagnosed at each of the units will be assessed for inclusion in the STAR pathway if suitable for EVAR. The study anticipates the assessment of over 200 AAA patients with the aim of recruiting up to 100 patients into the study to undergo EVAR using the STAR pathway.

Patients may be enrolled into the study to undergo EVAR using the STAR pathway provided all inclusion and no exclusion criteria are met. Subjects will be evaluated through to hospital discharge, receive a telephone call at 48 hours, return for follow-up visits at one month, and telephone follow-ups at three- and six months post treatment. Patients recruited into the study will have their routine clinical data collected at 12 months when they return for follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* They have been assessed as suitable for standard infrarenal EVAR within the manufacturer's "Instructions for Use" for the chosen endograft.
* Age over 55 (effectively excluding connective tissue disease)
* Fully independent at home or adequate provision for home care after discharge which would enable patients to perform basic activities of daily living including mobility, eating, drinking, and bathing
* Living with a partner or family member or having similar help available for the first 24-hours after discharge from the hospital
* Transport to attend the hospital in which they were treated within 1 hour for the first 24-hours after discharge. Should an ambulance not be readily available to attend the hospital within this timeframe, patients must be made aware and agree to make their own transport arrangements.
* Capable of complying with Protocol requirements, including follow-up
* An Informed Consent Form signed by the participant or legal representative

Exclusion Criteria:

* Significant cardiac disease, defined as one or more major predictors of increased perioperative cardiovascular risk according to the American College of Cardiology Cardiac Risk Classification, which remains untreated at the time of surgery
* Significant renal failure (pre-operative creatinine level of over 150 μmol/L or GFR less than 30mL/min/1.73m2 indicating severe chronic kidney disease (stage IV)
* Significant respiratory disease needing increased post-operative care not available in the home environment (e.g., nebulisers or oxygen therapy which is not set up at home)
* Any other condition, which in the opinion of the multidisciplinary team makes discharge within 23-hours unsafe
* Patients who lack capacity to consent to 23-hour EVAR will be excluded from the study
* There is concurrent enrolment in another drug or medical device study or have recently been involved in any research prior to recruitment

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with an infrarenal abdominal aortic aneurysm in at least five sites will be assessed for inclusion into the study. This is expected to be over 200 patients in five high-volume sites. From these patients, suitable patients will be able to be enrolled in the STAR pathway. The investigators expect approximately 100 patients to be enrolled from five UK centres.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Eligibility | 12 months
  Proportion of patients suitable for a short stay pathway (assessed in 200 patients)
Uptake | 12 months
  Proportion of patients who will accept admission to this pathway (assessed in all eligible patients)
Viability | 12 months
  Proportion of patients admitted to the short-stay pathway that can be discharged
  at 23-hours
Treatment satisfaction | 18 months
  Treatment satisfaction will be measured using the validated Aneurysm TSQ questionnaire
Patient well-being and stress | 18 months
  Well-being (W-B16) questionnaires will be used to measure depressed and anxious mood, energy, positive well-being, and stress at baseline, at 2-4 days and 30 days post-op
Quality of life measure | 18 months
  EQ-5D-5L health status questionnaires will be administered at baseline, 3- and 6-months post-op
Safety: Adverse events, readmissions and mortality | 24 months
  Rate of device-related and other adverse events, readmission, mortality (at 30, 90 days and 6- and 12- months) of patients
Costs up to 6 months | 18 months
  Inpatient micro-costing, surveys, as well as health resource use after discharged will be measured as any increase in social care and/or informal care

SECONDARY OUTCOMES:
Qualitative data | 12 months
  Describing the experiences, worries and concerns of patients, families and GPs as well as staff involved in the implementation of STAR, thus identifying the key barriers and drivers to implementation of a 23-hour pathway
Creation of a 'STAR tool-kit' | 12 months
  This may be used for implementation of a short-stay pathway in a wider group, to ensure sustainability. The toolkit will be produced if there are a significant proportion eligible and accepting the pathway and the pathway is viable without perceived safety issues

CONTACTS AND LOCATIONS:
Overall Officials: Colin Bicknell, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenhalgh RM, Brown LC, Kwong GP, Powell JT, Thompson SG; EVAR trial participants. Comparison of endovascular aneurysm repair with open repair in patients with abdominal aortic aneurysm (EVAR trial 1), 30-day operative mortality results: randomised controlled trial. Lancet. 2004 Sep 4-10;364(9437):843-8. doi: 10.1016/S0140-6736(04)16979-1. PMID 15351191
- [Background] Epstein D, Sculpher MJ, Powell JT, Thompson SG, Brown LC, Greenhalgh RM. Long-term cost-effectiveness analysis of endovascular versus open repair for abdominal aortic aneurysm based on four randomized clinical trials. Br J Surg. 2014 May;101(6):623-31. doi: 10.1002/bjs.9464. Epub 2014 Mar 24. PMID 24664537
- [Background] Brown LC, Powell JT, Thompson SG, Epstein DM, Sculpher MJ, Greenhalgh RM. The UK EndoVascular Aneurysm Repair (EVAR) trials: randomised trials of EVAR versus standard therapy. Health Technol Assess. 2012;16(9):1-218. doi: 10.3310/hta16090. PMID 22381040
- [Background] Shaw SE, Preece R, Stenson KM, De Bruin JL, Loftus IM, Holt PJE, Patterson BO. Short Stay EVAR is Safe and Cost Effective. Eur J Vasc Endovasc Surg. 2019 Mar;57(3):368-373. doi: 10.1016/j.ejvs.2018.10.008. Epub 2018 Nov 12. PMID 30442563
- [Background] Al-Zuhir N, Wong J, Nammuni I, Curran G, Tang T, Varty K. Selection, thirty day outcome and costs for short stay endovascular aortic aneurysm repair (SEVAR). Eur J Vasc Endovasc Surg. 2012 Jun;43(6):662-5. doi: 10.1016/j.ejvs.2012.02.031. Epub 2012 Mar 26. PMID 22456002
- [Background] Lachat ML, Pecoraro F, Mayer D, Guillet C, Glenck M, Rancic Z, Schmidt CA, Puippe G, Veith FJ, Bleyn J, Bettex D. Outpatient endovascular aortic aneurysm repair: experience in 100 consecutive patients. Ann Surg. 2013 Nov;258(5):754-8; discussion 758-9. doi: 10.1097/SLA.0b013e3182a617f1. PMID 24045449
- [Background] Krajcer Z, Ramaiah VG, Henao EA, Metzger DC, Nelson WK, Moursi MM, Rajasinghe HA, Al-Dallow R, Miller LE; LIFE Registry Investigators. Perioperative Outcomes From the Prospective Multicenter Least Invasive Fast-Track EVAR (LIFE) Registry. J Endovasc Ther. 2018 Feb;25(1):6-13. doi: 10.1177/1526602817747871. Epub 2017 Dec 18. PMID 29251207
- [Background] Block PC, Ockene I, Goldberg RJ, Butterly J, Block EH, Degon C, Beiser A, Colton T. A prospective randomized trial of outpatient versus inpatient cardiac catheterization. N Engl J Med. 1988 Nov 10;319(19):1251-5. doi: 10.1056/NEJM198811103191904. PMID 3185621
- [Background] Vaughan J, Gurusamy KS, Davidson BR. Day-surgery versus overnight stay surgery for laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2013 Jul 31;2013(7):CD006798. doi: 10.1002/14651858.CD006798.pub4. PMID 23904112
- [Background] Paton F, Chambers D, Wilson P, Eastwood A, Craig D, Fox D, Jayne D, McGinnes E. Initiatives to reduce length of stay in acute hospital settings: a rapid synthesis of evidence relating to enhanced recovery programmes. Southampton (UK): NIHR Journals Library; 2014 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK259855/ PMID 25642551
- [Background] Scantling-Birch Y, Martin G, Balaji S, Trant J, Nordon I, Malina M, Riga C, Bicknell C. Examining the impact of psychological distress on short-term postoperative outcomes after elective endovascular aneurysm repair (EVAR). J Psychosom Res. 2021 Mar;142:110367. doi: 10.1016/j.jpsychores.2021.110367. Epub 2021 Jan 19. PMID 33503514
- [Background] Dhesi J. Improving outcomes in older people undergoing elective surgery. J R Coll Physicians Edinb. 2010 Dec;40(4):348-53. doi: 10.4997/jrcpe.2010.416. PMID 21254711
- [Background] Romaine J, Peach G, Thompson M, Hinchliffe RJ, Bradley C. Psychometric validation of three new condition-specific questionnaires to assess quality of life, symptoms and treatment satisfaction of patients with aortic aneurysm. J Patient Rep Outcomes. 2019 May 16;3(1):29. doi: 10.1186/s41687-019-0119-0. PMID 31098754
- [Background] Peach G, Romaine J, Wilson A, Holt PJ, Thompson MM, Hinchliffe RJ, Bradley C. Design of new patient-reported outcome measures to assess quality of life, symptoms and treatment satisfaction in patients with abdominal aortic aneurysm. Br J Surg. 2016 Jul;103(8):1003-11. doi: 10.1002/bjs.10181. Epub 2016 May 23. PMID 27214517
- [Background] Fleisher LA, Beckman JA, Brown KA, Calkins H, Chaikof E, Fleischmann KE, Freeman WK, Froehlich JB, Kasper EK, Kersten JR, Riegel B, Robb JF, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Buller CE, Creager MA, Ettinger SM, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Hunt SA, Lytle BW, Nishimura R, Ornato JP, Page RL, Tarkington LG, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines on Perioperative Cardiovascular Evaluation for Noncardiac Surgery); American Society of Echocardiography; American Society of Nuclear Cardiology; Heart Rhythm Society; Society of Cardiovascular Anesthesiologists; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society for Vascular Surgery. ACC/AHA 2007 guidelines on perioperative cardiovascular evaluation and care for noncardiac surgery: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines on Perioperative Cardiovascular Evaluation for Noncardiac Surgery): developed in collaboration with the American Society of Echocardiography, American Society of Nuclear Cardiology, Heart Rhythm Society, Society of Cardiovascular Anesthesiologists, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, and Society for Vascular Surgery. Circulation. 2007 Oct 23;116(17):e418-99. doi: 10.1161/CIRCULATIONAHA.107.185699. Epub 2007 Sep 27. No abstract available. PMID 17901357
- [Background] Hlatky MA, Boineau RE, Higginbotham MB, Lee KL, Mark DB, Califf RM, Cobb FR, Pryor DB. A brief self-administered questionnaire to determine functional capacity (the Duke Activity Status Index). Am J Cardiol. 1989 Sep 15;64(10):651-4. doi: 10.1016/0002-9149(89)90496-7. PMID 2782256
- See also: The NHS Outcomes Framework 2013/14 — https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment_data/file/213055/121109-NHS-Outcomes-Framework-2013-14.pdf
- See also: Enhanced recovery care pathway: A better journey for patients seven days a week and better deal for the NHS — https://www.stgeorges.nhs.uk/wp-content/uploads/2015/01/ERP-care-pathway-A-better-journey-for-patients-seven-days-a-week-and-better-deal-for-the-NHS.pdf